CLINICAL TRIAL: NCT04897789
Title: The Early Head Start Family and Child Experiences Survey (Baby FACES 2018)
Acronym: BabyFACES18
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Office of Planning, Research & Evaluation (U.S. Federal Agency); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 50193
Record Dates: First submitted 2021-05-17; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Early Head Start Participation
Keywords: child care; child development; child health; child nutrition; child rearing; children; early childhood education; Early Head Start; families; parenting skills; parents; relationships

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- children/pregnant women: children/pregnant women (2,310)
- parents: parents (2,310)
- classrooms/teachers: classrooms/teachers (840)
- home visitors: home visitors (630)
- center directors: center directors (493)
- program directors: program directors (140)

SUMMARY:
Early Head Start (EHS) Family and Child Experiences Survey - 2018 (Baby FACES 2018) will answer new questions about EHS programs, staff, and families that can guide program technical assistance, management, and policy. It will provide information about EHS programs in the context of the adoption of the new Head Start Early Learning Outcomes Framework. Baby FACES 2018 will consist of two nationally representative cross-sectional samples of programs, centers, classrooms, home visitors, and children and families. It will include surveys of program directors, center directors, teachers, home visitors, and parents; conduct observations of classrooms and home visits, and ask staff and parents to report on children's development.

DETAILED DESCRIPTION:
The overarching purpose of the Baby FACES studies is to provide knowledge about Early Head Start children and families, and the EHS programs and staff who serve them. The ongoing series of Baby FACES data collections is aimed at maintaining up-to-date core information on EHS over time while also focusing on different areas of interest. The Baby FACES studies began with Baby FACES 2009, a longitudinal descriptive study that followed two cohorts of children and families through participation in the program and focused on program services and participation, and child and family wellbeing and outcomes over time. Baby FACES 2018 (and a future round in 2022) have been redesigned to provide cross-sectional descriptive information and a point in time picture of EHS. The present study will focus on understanding the processes in EHS core services (classrooms and home visits) that support infant and toddler development; namely, nurturing and responsive relationships between children and caregivers. With this new focus, Baby FACES 2018 will take a more in depth look at classrooms while a future study, Baby FACES 2022, will take a more in depth look at home visiting.

The Baby FACES team will carry out a descriptive study that includes a nationally representative sample of EHS programs, centers, classrooms, teachers, home visitors, and children and families (including pregnant women) and answers new questions about how EHS programs function. The study is guided by a comprehensive conceptual framework that illustrates how EHS program processes and activities are expected to lead to high quality service delivery and enhanced family and infant/toddler outcomes for the program overall. The overarching research question for Baby FACES 2018 is: How do EHS services support infant/toddler growth and development in the context of nurturing, responsive relationships? The study will address this question through the collection of rich information using interviews, self-administered questionnaires, classroom observations, and administrative data sources. This approach will allow the Administration for Children and Families to capture important information about EHS services, families, and children across all service options (e.g., center-based, home-based, or those providing both service options), as well as in depth information about how EHS classrooms and teacher-child relationships support infant/toddler development.

ELIGIBILITY:
Inclusion Criteria:

* The Early Head Start programs participating in Baby FACES 2018 are a probability sample selected from among study-eligible programs on the 2016-2017 Head Start Program Information Report (PIR). To be eligible for the study, a program had to be
* In one of the 50 states or the District of Columbia
* Providing services directly to pregnant women or children up to preschool age.
* Not be in imminent danger of losing its grantee status.

Exclusion Criteria:

* American Indian and Alaska Native Head Start programs (Region XI) or Migrant and Seasonal Worker Head Start programs (Region XII) were not eligible.

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Early Head Start pregnant women and Early Heat Start infants and toddlers (and their families), Early Head Start programs, Early Head Start centers, Early Head Start home visitors, Early Head Start classrooms/teachers
Sampling Method: Probability Sample
Enrollment: 6723 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Classroom quality/teacher-child interactions | One-day observation in March-May 2018
  Indicators of classroom quality were assessed using the Classroom Assessment Scoring System, Infant version (CLASS-I), depending on the ages of children in the classroom. The CLASS assesses the quality of interactions between teachers and children in classrooms. Please see the Baby FACES User's Manual (Cannon et al. 2020) for more information on scores and technical properties.
Classroom quality/teacher-child interactions | One-day observation in March-May 2018
  Indicators of classroom quality were assessed using the Classroom Assessment Scoring System, Toddler version (CLASS-T), depending on the ages of children in the classroom. The CLASS assesses the quality of interactions between teachers and children in classrooms. Please see the Baby FACES User's Manual (Cannon et al. 2020) for more information on scores and technical properties.
Classroom quality/teacher-child interactions | One-day observation in March-May 2018
  Indicators of classroom quality were assessed using the Quality of Caregiver Child Interactions for Infants and Toddlers (Q-CCIIT). The Q-CCIIT assesses the quality of interactions between teachers and children in classrooms. Please see the Baby FACES User's Manual (Cannon et al. 2020) for more information on scores and technical properties.
Child expressive and receptive vocabulary | 1 week
  Teachers and parents independently reported on words the child understands and says, using the MacArthur Communicative Development Inventories (CDI). Please see the Baby FACES User's Manual (Cannon et al. 2020) for more information on scores and technical properties.
Child social-emotional/behavioral development | 1 week
  Teachers and parents independently reported on children's social competence and problem behaviors using the Brief Infant Toddler Social Emotional Assessment. Please see the Baby FACES User's Manual (Cannon et al. 2020) for more information on scores and technical properties.

SECONDARY OUTCOMES:
Teacher-child relationships | 1 week
  Teachers report on their relationship with children using the Student-Teacher Relationship, Short Form. Please see the Baby FACES 2018 User's Manual (Cannon et al. 2020) for more information on the scores and technical properties.
Parent-child relationships | 1 week
  Parent-child relationships were assessed with the Child-Parent Relationship Scale, Short Form. Please see the Baby FACES 2018 User's Manual (Cannon et al. 2020) for more information on the scores and technical properties.
Parent-child relationships | 1 week
  Parent-child relationships were assessed with the Healthy Families Parenting Inventory. Please see the Baby FACES 2018 User's Manual (Cannon et al. 2020) for more information on the scores and technical properties.

CONTACTS AND LOCATIONS:
Overall Officials: Cheri Vogel, Ph.D., Study Director — Mathematica Policy Research; Sally Atkins-Burnett, Ph.D., Principal Investigator — Mathematica Policy Research; Yange Xue, Ph.D., Principal Investigator — Mathematica Policy Research
Locations (1):
- Mathematica Policy Research, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
In the future, Baby FACES archived data will be available for access
Time Frame: Data will become available within 2 years of the completion of each study wave.
Access Criteria: Applications for access to restricted-use data file include completing and adhering to a User Agreement.